CLINICAL TRIAL: NCT02919462
Title: Open-label, Multicenter, Randomized Phase II Trial of Treatment With Cisplatin and Pemetrexed or Cisplatin and Oral Vinorelbine in Chemotherapy Naïve Patients Affected by Stage IIIB-IV Non-Squamous Non-Small Cell Lung Cancer With High Thymidylate Synthase Expression
Acronym: HighTySy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitement rate
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST162.10; 2015-003440-39 (EudraCT Number)
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Secondary; Advanced Stage IIIB; High Thymidylate Synthase Expression
Keywords: Carcinoma, Non-Small-Cell Lung; advanced stage IIIB; high Thymidylate Synthase expression; Treatment; Chemotherapy Naïve Patients; stage IIIB-IV Non-Squamous Non-Small Cell Lung Cancer; Cisplatin and Pemetrexed; Cisplatin and Oral Vinorelbine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Vinorelbine; Cisplatin; Maintenance; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A (Experimental): Oral vinorelbine 60-80 mg/m2 on days 1 and 8 (first cycle 60 mg/m2) + Cisplatin 80 mg/m2 on day 1 every 3 weeks, for 4 cycles.
  Maintenance with Metronomic Oral Vinorelbine 50 mg three times a week on Monday, Wednesday and Friday continuously until disease progression, patient refusal or excessive toxicity (1 cycle: 3 weeks).
  Interventions: Drug: Oral vinorelbine; Drug: Cisplatin; Drug: Maintenance with Metronomic Oral Vinorelbine
- Treatment Arm B (Active Comparator): Pemetrexed, 500 mg/m2, day 1 + Cisplatin, 75 mg/m2, day 1 every 3 weeks, for 4 cycles.
  Maintenance with Pemetrexed 500 mg/m2 day1 q 21 until disease progression (1 cycle: 3 weeks).
  7-10 days before treatment administration, premedication with vitamin B12 1000µg intramuscular injection (every 9 weeks) and folate 1mg every day should be commenced.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Maintenance with Pemetrexed

INTERVENTIONS:
Drug: Oral vinorelbine — Oral vinorelbine 60-80 mg/m2 on days 1 and 8 (first cycle 60 mg/m2) every 3 weeks, for 4 cycles
  Arms: Treatment Arm A
Drug: Cisplatin — Cisplatin 80 mg/m2 on day 1 every 3 weeks, for 4 cycles
  Arms: Treatment Arm A
Drug: Maintenance with Metronomic Oral Vinorelbine — Maintenance with Metronomic Oral Vinorelbine 50 mg three times a week on Monday, Wednesday and Friday continuously until disease progression, patient refusal or excessive toxicity (1 cycle: 3 weeks).
  Arms: Treatment Arm A
Drug: Pemetrexed — Pemetrexed, 500 mg/m2, day 1 every 3 weeks, for 4 cycles
  Arms: Treatment Arm B
Drug: Cisplatin — Cisplatin 75 mg/m2, day 1 every 3 weeks, for 4 cycles
  Arms: Treatment Arm B
Drug: Maintenance with Pemetrexed — Maintenance with Pemetrexed 500 mg/m2 day1 q 21 until disease progression (1 cycle: 3 weeks)
  Arms: Treatment Arm B

SUMMARY:
This is an open-label, multicentre, randomized phase II trial.

Eligible patients with Non Small Cell Lung Cancer (NSCLC) with high Thymidylate Synthase (TS) expression , will be randomly assigned with 1:1 ratio to the following treatment Arms:

A. 4 cycles of Cisplatin + Oral Vinorelbine followed by maintenance with Metronomic Oral Vinorelbine until disease progression

B. 4 cycles of Cisplatin + Pemetrexed followed by maintenance with Pemetrexed until disease progression

Treatment will be repeated every 21 days .

DETAILED DESCRIPTION:
An Open-label, Multicenter, Randomized Phase II Trial of Treatment with Cisplatin and Pemetrexed or Cisplatin and Oral Vinorelbine in Chemotherapy Naïve Patients affected by stage IIIB-IV Non-Squamous Non-Small Cell Lung Cancer with high Thymidylate Synthase (TS)expression After signing the informed consent for TS expression evaluation (see Appendix A), patients will be tested for TS expression status of their tumor tissue.

If TS expression is more than 70 in the nucleus or ≥210 in nucleus and in the cytoplasm of tumor cell, they will be categorized as high TS expression patients, and if it is less, they will be considered as TS-negative.

Study Treatment:

Eligible patients will be randomly assigned to the following treatment Arms:

A. Oral vinorelbine 60-80 mg/m2 on days 1 and 8 (first cycle 60 mg/m2) + Cisplatin 80 mg/m2 on day 1 every 3 weeks, for 4 cycles.

Maintenance with Metronomic Oral Vinorelbine 50 mg three times a week on Monday, Wednesday and Friday continuously until disease progression, patient refusal or excessive toxicity (1 cycle: 3 weeks).

B. Pemetrexed, 500 mg/m2, day 1 + Cisplatin, 75 mg/m2, day 1 every 3 weeks, for 4 cycles.

Maintenance with Pemetrexed 500 mg/m2 day1 q 21 until disease progression (1 cycle: 3 weeks).

7-10 days before treatment administration, premedication with vitamin B12 1000µg intramuscular injection (every 9 weeks) and folate 1mg every day should be commenced.

The total duration of the study will be 3 years. The enrollment period wil be 2 years and 1 year of follow up. Treatment period: until disease progression, intolerable toxicity or patient refusal.

Number of Subjects :130 patients (65 patients per arm)

Statistical Methodology The primary variable of this study is Disease Control Rate (DCR). According to primary variable, assuming a DCR≥70% for patients with high TS expression treated with cisplatin and vinorelbine and a DCR=44% for patients with high TS expression treated with cisplatin and pemetrexed, considering a 2-tailed alpha=0.05 and beta=0.10, it is necessary to enroll 65 patients per arm (130 patients in total) in a 24-month period and the subsequent 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically Non-squamous NSCLC, (including those with a non-specified tumor type).
2. Metastatic (stage IV, both M1A or M1B) or locally advanced (stage IIIB, with metastasis to supraclavicular nodes) according to TNM VII edition.
3. TS nuclear H-score ≥ 70 or with TS nuclear and cytoplasmatic H-score ≥ 210.
4. Patients at first diagnosis or those with disease recurrence after former surgery are eligible.
5. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan. See section 9.2 and Appendix E for the evaluation of measurable disease.
6. At least one target or non-target lesion not previously irradiated according to RECIST version 1.1
7. Male or Female, aged ≥18 years.
8. Life expectancy greater than 3 months.
9. ECOG performance status ≤2 (see Appendix C).
10. Patients must have normal organ and marrow function as defined below:

    * leukocytes ≥3,000/µL
    * absolute neutrophil count ≥1,000µL
    * platelets ≥100,000/µL
    * total bilirubin within normal institutional limits
    * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
    * creatinine within normal institutional limits OR
    * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
11. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
12. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Prior chemotherapy or therapy with systemic anti-neoplastic therapy for advanced disease.
2. Prior surgery and/or localised irradiation is permitted if delivered outside to the target lesion.
3. Prior adjuvant chemotherapy is permitted if it did not contain vinorelbine and pemetrexed and if administered at least 6 months prior entering the study.
4. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
5. Patients with symptomatic brain metastasis or spinal cord compression that has not yet been treated with surgery and/or radiation. Patients with CNS metastases or spinal cord compression previously treated with surgery and/or radiation are eligible if they are asymptomatic and do not require escalating high dose steroids (anti-seizure medications are allowed)
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to pemetrexed, vinorelbine, cisplatin, carboplatin or other agents used in the study.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix or surgically resected prostate cancer with normal PSA);
9. NSCLC with EGFR mutation (or not able to use EGFR inhibitor) or with anaplastic lymphoma kinase (ALK) gene translocation (such as EML4-ALK).
10. Has a known allergy, hypersensitivity, or contraindication to cisplatin, pemetrexed, or vinorelbine or any components used in their preparation or has a contraindication specified in section 7.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | up to 36 months
  Rate (DCR; complete response (CR) plus partial response (PR) plus stable disease (SD)). The response is assessed according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Toxicity | up to 36 months
  Toxicity assessed after each cycle using the Common Toxicity Criteria AE (version 4.03)
Overall survival (OS) within th 2 arms | up to 36 months
  Overall Survival (OS) is defined as the observed length of life from study entry to death for any cause or the date of last contact for patients lost to follow up
Progression free survival (PFS) within the two arms | up to 36 months
  Progression free survival (PFS) is the time from the date of randomization to the date of the first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
optimal TS H-score cutpoint | up to 36 months
  to define the optimal Thymidylate Synthase expression(TS) H-score cutpoint in cytoplasm and/or nucleus . TS nuclear and cytoplasmic staining will be evaluated by using an intensity scale (0-3) and the percentage of cells in each category, resulting in semiquantitative H scores ranging from 0 to 300 will be calculated. Total TS H-scores will be calculated posthoc as the sum of nuclear and cytoplasm TS H-scores (range 0-600).

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Dazzi, MD, Principal Investigator — UOC Oncologia Medica - PO di Ravenna - AUSL della Romagna-RAVENNA Viale Randi 5 - 48121 Ravenna
Locations (5):
- Italy (5):
  - Ircc Irst, Meldola, FC
  - U.O. Oncologia Medica, Faenza, RA
  - Claudio Dazzi, Ravenna, RA
  - Ospedale di Piacenza, ASL Piacenza, Piacenza
  - U.O. Oncologia Ospedale degli Infermi, Rimini

IPD SHARING:
Plan to Share IPD: Undecided